CLINICAL TRIAL: NCT04673058
Title: Effectiveness of Spinal Manipulation in Addition to Standard Pharmacological Treatment in Fibromyalgia : A Blinded Randomized Clinical Trial
Brief Title: Effectiveness of Spinal Manipulation in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Bugra Ince, MD Bugra Ince, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BI031220
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; manipulation; manual therapy; spinal
MeSH Terms: conditions — Fibromyalgia | interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: Prospective, triple-blinding, randomized controlled and 3-arm parallel group design clinical study. 3 arms of the study were planned to consist of active intervention group, sham treatment group and no intervention group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 2 staff members who will administer the treatment to active intervention and sham therapy groups will not be able to be blinded due the inherent of manual therapy. Staff members who are responsible for statistical analysis, participants and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal Manipulation Group (Experimental): After the patients were evaluated in terms of somatic dysfunction, the appropriate techniques of Cervical Upglide Thrust, Cervical Downglide Thrust, Cervical Traction Thrust, Cervical Rotation Thrust, Cervico-Thoracic Distraction Manipulation, Cervico-Thoracic Lateral Glide (Spinous Push) Manipulation, Supine Screw Thoracic Thrust, Prone Thoracic Thrust, and Lumbar Spine Rotation Manipulation will be applied to patients.
  Interventions: Procedure: Spinal Manipulation
- Sham Manipulation Group (Sham Comparator): A treatment will be applied which is very similar to active treatment but aimed to have minimal therapeutic effect. For this, the practitioner will primarily identify the areas where somatic dysfunction is detected and keep the application away from these areas. The patient will be positioned for treatment as in active therapy, but once in the lock position, a lower thrust will be given by releasing some back from the position. In this way, the movement will be imitated without reaching the elastic zone and a stronger similarity will be provided compared to sham treatments such as light touch or massage.
  Interventions: Procedure: Sham Manipulation
- No Intervention Group (No Intervention): These patients will receive only their pharmacological treatments.

INTERVENTIONS:
Procedure: Spinal Manipulation — Intervention will be administered twice a week for 3 weeks. Each treatment session will be given in 20-minute sessions consisting of 10 minutes of manual examination and 10 minutes of manual treatment.
  Other Names: high velocity low amplitude thrust manipulation
  Arms: Spinal Manipulation Group
Procedure: Sham Manipulation — The practitioner will primarily identify the areas where somatic dysfunction is detected and keep the application away from these areas. The patient will be positioned for treatment as in active therapy, but once in the lock position, a lower thrust will be given by releasing some back from the position.
  Arms: Sham Manipulation Group

SUMMARY:
The aim of this study is to evaluate whether spinal manipulation, which is a potential treatment method for musculoskeletal pain, has an additional contribution in patients with fibromyalgia receiving standard pharmacological treatment.

DETAILED DESCRIPTION:
Although fibromyalgia (FM) is quite common, success rates in conservative treatment are unsatisfying. Combination of pharmacological and non-pharmacological applications is recommended in treatment. Although the etiology of FM is not well known, characteristic findings such as hyperalgesia and allodynia suggest problems related to pain and sensorial processing in the central nervous system.

It has been suggested that spinal manipulation can alter sensorimotor integration in the central nervous system and therefore can be used in the treatment of central sensitization syndromes. However, manual therapy applications, which were examined under the heading of chiropractic in the 2016 EULAR treatment recommendations, were not recommended due to the low quality (open-label, quasi-experimental) of the studies conducted so far. However, it has been suggested for future studies to investigate whether the combined use of pharmacological and non-pharmacological treatments is more effective than single modality management. But since then unfortunately a high level of evidence also could not be obtained related to use of spinal manipulation in FM due to reasons such as lack of reporting of the manual therapy methods used in detail, conducting studies involving mostly soft tissue techniques and not following CONSORT recommendations.

This study is planned as a prospective, triple-blinding, randomized controlled and 3-arm parallel group design clinical study considering the concepts that have been lacking the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with fibromyalgia according to the 2016 ACR Fibromyalgia Diagnostic Criteria
* Having been receiving pharmacological treatment for fibromyalgia for at least 2 weeks
* VAS pain score> 4

Exclusion Criteria:

* Structural problem of the musculoskeletal system (acute spinal disc herniation, acute spondylolisthesis / lysis, fractures and dislocations, advanced degenerative changes, spinal stenosis)
* Pregnancy or breastfeeding
* Inflammatory or infectious disease
* Malignancy
* Neuromuscular disease
* History of spinal surgery
* Unstable psychiatric disease
* Previously received manual therapy or having enough information about manual therapy to distinguish between sham and real therapy (researched online, watched videos…).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female Patients
Enrollment: 60 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain Intensity at 1 and 3 months | Baseline, one week after the last treatment session (1st month) and 3rd month
  Patients will be asked to mark their pain on the visual analog scale (VAS) during each visits.

SECONDARY OUTCOMES:
Change from Baseline Tenderness (tender point pain threshold score) at 1 and 3 months | Baseline, one week after the last treatment session (1st month) and 3rd month
  Pressure pain threshold of 18 points specified in 1990 American Collage of Rheumatology (ACR) Fibromyalgia classification criteria will be evaluated with The Lafayette Manual Muscle Tester Model 01165 (Lafayette Instrument Company, Lafayette IN, USA). This device is a dynamometer. It has been shown that if circumference is used instead of area as the correction coefficient hand dynamometers with wider tips than standard algometers are also valid and reliable in the pressure pain threshold measurement. The Lafayette Hand-Held Dynamometer uses a tip with a circumference of 5.65 cm. The applied force (kg) / 5.65 will be used as the pressure pain threshold unit in the study. The arithmetic mean of the data obtained from 18 points will be recorded as the tender point pain threshold score.
Change from Baseline Revised Fibromyalgia Impact Questionnaire (FIQR) at 1 and 3 months | Baseline, one week after the last treatment session (1st month) and 3rd month
  FIQR consists of 3 domains. The first domain contains 9 questions that can be scored between 0 and 10 and the score of the physical function is found by dividing the total score by three. Second domain contains 2 questions and the overall impact score is the sum of the scores from these two questions. Third domain consists of 10 questions and symptom score is obtained by dividing the total score by two. Total FIQR score is the sum of 3 domain points.
Change from Baseline Pain Extent at 1 and 3 months | Baseline, one week after the last treatment session (1st month) and 3rd month
  The extent of the pain will be evaluated by widespread pain index (WPI). The WPI quantifies the extent of bodily pain on a 0-19 scale by asking patients if they have had pain or tenderness in 19 different body regions (shoulder girdle, hip, jaw, upper arm, upper leg, lower arm, and lower leg on each side of the body, as well as upper back, lower back, chest, neck, and abdomen) over the past week, with each painful or tender region scoring 1 point.
Change from Baseline Fibromyalgia Severity Score (FSS) at 1 and 3 months | Baseline, one week after the last treatment session (1st month) and 3rd month
  FSS is the sum of the WPI and symptom severity scale (SSS) scores. SSS consists of two domains. For the first domain, the complaints of fatigue, waking unrefreshed and cognitive symptoms are scored between 0 (no problem) and 3 (life-disturbing problems
  ). For the second domain, headaches, pain or cramps in lower abdomen, and depression are scored between 0 (absent) and 1 (present). The total score gives the SSS score.

CONTACTS AND LOCATIONS:
Overall Officials: Bugra Ince, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing will be done on request.

REFERENCES:
- [Background] Haavik-Taylor H, Murphy B. Cervical spine manipulation alters sensorimotor integration: a somatosensory evoked potential study. Clin Neurophysiol. 2007 Feb;118(2):391-402. doi: 10.1016/j.clinph.2006.09.014. Epub 2006 Nov 29. PMID 17137836
- [Background] Moustafa IM, Diab AA. The addition of upper cervical manipulative therapy in the treatment of patients with fibromyalgia: a randomized controlled trial. Rheumatol Int. 2015 Jul;35(7):1163-74. doi: 10.1007/s00296-015-3248-7. Epub 2015 Mar 18. PMID 25782585
- [Background] Haller H, Lauche R, Sundberg T, Dobos G, Cramer H. Craniosacral therapy for chronic pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2019 Dec 31;21(1):1. doi: 10.1186/s12891-019-3017-y. PMID 31892357
- [Background] Licciardone JC, Brimhall AK, King LN. Osteopathic manipulative treatment for low back pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2005 Aug 4;6:43. doi: 10.1186/1471-2474-6-43. PMID 16080794
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Derived] Ince B, Kara M, Erdem I, Yurdakul OV, Erden T, Aydin T. Effectiveness of spinal manipulation in addition to pharmacological treatment in fibromyalgia: A blinded randomized trial. PM R. 2023 Mar;15(3):342-351. doi: 10.1002/pmrj.12953. Epub 2023 Feb 16. PMID 36695286